CLINICAL TRIAL: NCT05083273
Title: Life Experience of People Aged 60 and Over Living with HIV: Quantitative Sociological Study
Brief Title: Life Experience of People Aged 60 and Over Living with HIV
Acronym: PVVIH
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1321
Record Dates: First submitted 2021-06-01; First posted 2021-10-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-06

CONDITIONS: Virus-HIV
Keywords: VIH; Living with HIV; 60 years old and over
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Cohorte — Completion of a socio-demographic, professional, medical and personal questionnaire
  Other Names: Questionnaire

SUMMARY:
The purpose of this study is to Assess the impact of HIV on the life course of patients aged 60 and over.

DETAILED DESCRIPTION:
COREVIH IDF Nord and CERMES3 conducted a first qualitative survey of 32 HIV patients aged 60 and over. The study, in the form of an individual interview, aimed to identify the difficulties that PLWHIV may encounter in their life course, to question their future and the impact that HIV could have.

From this study, a questionnaire was drawn up covering the points raised by the qualitative study. The questionnaire was designed by doctors of the four hospitals that participated in the first study and a sociologist from CERMES3.

After patient's oral agreement obtained, the study questionnaire "Sociological study PVHIV ≥ 60 years" will be given to the patient for completion.

ELIGIBILITY:
Inclusion Criteria :

People aged 60 and over living with HIV and view in consultation

Patient participation agreement obtained

Exclusion criteria :

People living with HIV less than 60 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged 60 and over living with HIV
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Determine the impact of HIV in the life cours of people aged 60 and over and the questioning of the future. | Through study completion, an average of 6 month
  People aged 60 and over will answer to a sociological questionnaire to identify the impact of HIV in their life cours and the questioning of the future, directly or indirectly linked to HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Blum, Dr, Principal Investigator — Hôpital NOVO
Locations (6):
- France (6):
  - Hospital Beaujon, Clichy / Médecine Interne, Clichy
  - Université Paris Descartes - CERMES3, Paris
  - Hôpital Bichat Claude-Bernard - Service de Maladies Infectieuses et Tropicales, Paris
  - Hôpital Bichat Claude-Bernard -COREVIH Ile de France Nord, Paris
  - Centre Hospitalier René Dubos, Pontoise
  - Hospital Delafontaine, Saint-Denis / Maladie infectieuse, Saint-Denis